CLINICAL TRIAL: NCT02538874
Title: A Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986171 in Healthy Subjects
Brief Title: A Study of BMS-986171 in Healthy People to Assess Safety, to Measure Blood Levels of Drug, and to Find Out What the Drug Does to the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MB007-005
Record Dates: First submitted 2015-08-21; First posted 2015-09-02 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Liver Fibrosis/NASH

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (Experimental): BMS-986171 or Placebo on specified days
  Interventions: Drug: BMS-986171; Other: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): BMS-986171 or Placebo on specified days
  Interventions: Drug: BMS-986171; Other: Placebo
- Part C: Multiple Ascending Dose in Japanese subjects (J-MAD) (Experimental): BMS-986171 or Placebo on specified days
  Interventions: Drug: BMS-986171; Other: Placebo

INTERVENTIONS:
Drug: BMS-986171
Other: Placebo

SUMMARY:
The purpose of this study is to assess safety, to measure blood levels of drug, and to find out what the drug does to the body.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Age 21 to 55 years (Part A,B, and C)
* BMI 30-40 (Part A or Part B); BMI 20-35 (Part C). BMI = weight (kg)/ [height (m)]

Exclusion Criteria:

* Any significant medical illness
* Cannot tolerate subcutaneous injections, or having blood samples taken
* Smoking more than 10 cigarettes/day
* History of allergy to pegylated compounds or of hypersensitivity to protein based therapeutics.
* HIV, Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection.
* Pregnancy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose of BMS-986171 will be measured by number of incidence of AEs, serious AEs, and events of special interest including injection site assessment, AEs leading to discontinuation | up to 30 days after the last dose
  Adverse Event (AE)
Safety and tolerability of multiple subcutaneous doses of BMS-986171 will be measured by number of incidence of AEs, serious AEs, and events of special interest including injection site assessment, AEs leading to discontinuation | up to 30 days after the last dose
Safety and tolerability of single dose of BMS-986171 will be measured by number of incidence of Death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to 30 days after the last dose
Safety and tolerability of multiple subcutaneous doses of BMS-986171 will be measured by number of incidence of Death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, physical examinations | up to 30 days after the last dose

SECONDARY OUTCOMES:
Immunogenicity based on antibody responses | 6 months following study discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Profil Institute For Clinical Research, Inc., Chula Vista, California
  - Wcct Global, Llc, Cypress, California

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx